CLINICAL TRIAL: NCT05607849
Title: Shared Decision-making for Breast Cancer Screening in Primary Care
Brief Title: Breast Cancer Screening Uptake: a Randomized Controlled Trial Assessing the Effect of a Decisional Aid
Acronym: DEDICACES2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: National Cancer Institute, France (Other Government); Nantes University hospital, Research Department (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC20_0532; 2024-A00987-40 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2022-10-24; First posted 2022-11-07 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer screening; Organized screening; General practitioner; Randomized controlled trial; Shared medical decision-making; Decisional aid; Primary health care
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decisional aid for organised cancer screening (Experimental): Women will receive a leaflet that presents the tool. The leaflet includes a link to access the tool, and encourages the person to consult their GP to initiate the shared decision-making process. GPs will receive a letter presenting the study that includes: a) information about shared decision-making and how to implement it; b) the letter that is sent to their patients, and c) a recommendation to implement shared decision-making with their patients.
  Interventions: Other: The decidons ensemble (let's decide together) leaflet and the discutons-mammo.fr (let's talk about breast cancer screening) online tool.
- Standard organised cancer screening (No Intervention): Women and their GPs will continue to carry out usual screening.

INTERVENTIONS:
Other: The decidons ensemble (let's decide together) leaflet and the discutons-mammo.fr (let's talk about breast cancer screening) online tool. — The leaflet will include a link to access the discutons-mammo.fr DA aid tool, and will inform women about shared decision-making.
  The GPs of women who are sent the leaflet will also be sent a letter encouraging shared decision-making. This material will be sent 3 months after women have received their breast cancer screening invitation letter.
  Data related to primary and secondary objectives will be collected by questionnaire from the 2 groups. The questionnaire will be sent 2 months after participants are informed about the tool.
  Arms: Decisional aid for organised cancer screening

SUMMARY:
Shared decision-making for organised breast cancer screening (OBCS) could be improved by fostering interaction and exchanges of information between women and General Practitioners (GPs), for instance by including an assistance tool in the dispatch of the invitation letter for Organised Screening for breast cancer. In 2018 the national cancer Institute funded the development of a decisional aid (DA) on the theme of whether or not to take part in breast cancer screening, specific to the French setting. It is the website Discutons-mammo.fr DEDICACES project 1.

DEDICACES 2 is a population-based trial with a cluster design. It studies humans, without modifying their usual care. The experiment assesses the effect of the discutons-mammo.fr tool on the decision to take part (or not) in OBCS among women who are invited for screening.

ELIGIBILITY:
Inclusion Criteria :

- General practitioners (GPs):

The following GPs will be included:

1) Practicing in one of the French départements (administrative area) covered by the study.

- Women:

The following women will be included:

1. Invited to participate in OBCS by the National Health Insurance Agency (Caisse Nationale d'Assurance Maladie; CNAM) during the studied month: eligible for OBCS, therefore aged between 50 and 74 at the time of inclusion;
2. On the patient list of a GP who is covered by the study at the time of inclusion;
3. Covered by one of the CPAM (Caisse Primaire d'Assurance Maladie) in the participating departments.

Exclusion Criteria :

- General practitioners (GPs) :

The following GPs will be excluded:

1. Those who do not have any patients invited for OBCS in the studied month;
2. Those whose practice does not correspond to the usual activities of a GP (known as a Mode d'Exercice Particulier), or who have very few patients (who have seen fewer than 100 different patients in the year preceding the experiment);
3. Those who practice within a health centre (as it is impossible to evaluate the activity of an individual practitioner in health insurance databases);
4. Those who explicitly state that they do not want to take part in the study, in response to an initial letter of invitation. This letter will inform them that the study is being run, and will inform them of the option to refuse to participate if they so wish;
5. Those who are participating in the MyPEBS study (the only national study of OBCS at the time the present protocol was drawn up).

   * Women:

The following women will not be included:

1. Participants in the MyPEBS study ( the only national study of OBCS at the time the present protocol was drawn up); or,
2. If their GP refuses to participate in the study; or,
3. women under guardianship.

The following women will be excluded:

* Those who object to the study in accordance with regulatory procedures issued by the Data Protection Officer (DPO),
* Those who do not respond within 1 month after the questionnaire has been sent.

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of the discutons-mammo.fr DA tool on decision-making concerning the choice of whether or not to participate in OBCS among women who are invited for screening. | 2 months
  Overall score on the 16-item Decisional Conflict Scale (DCS). Measured 2 months after participants are informed about the tool, in both arms. 5 response categories: 1 = strongly agree; 5 = strongly disagree. Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict].

SECONDARY OUTCOMES:
Evaluation of the effect of the presentation of the discutons-mammo.fr tool on the intention to participate in OBCS. | 2 months
  Score on a one-item (Measures of Decision) scale measuring intention to participate in OBCS. Measured 2 months after participants are informed about the tool, in both arms. Respondents check a box lying on a 15-point scale ranging from "I wish to participate in breast cancer screening" to "I do not wish to participate in breast cancer screening", with "I'm not sure" in the middle. Scores will be reclassified as follows: 1-5 (yes); 6-10 (unsure); 11-15 (no).
Evaluation of the effect of presenting the discutons-mammo.fr DA tool on the implementation of shared decision-making. | 2 months
  Scores on the 9-item Shared Decision Making Questionnaire (SDM Q9). Measured 2 months after presentation of the tool, in both arms. Six response categories: 10 = completely disagree; 5 = completely agree. Scores are reported on a scale ranging from 0 (the lowest possible level of SDM) to 100 ( the highest extent of SDM).
Evaluation of the effect of presenting the discutons-mammo.fr DA tool on women's knowledge of OBCS. | 2 months
  Number of correct responses to a 10-item questionnaire that tests OSBC-related knowledge. The questionnaire was developed in the context of the DEDICACES project (part 1) and is based on items included in the IPDAS (International Patient Decision Aid Standards) score. Measured 2 months after presentation of the support tool, in both arms.
Evaluation of the effect of the presentation of the discutons-mammo.fr DA tool on women's care pathways following an invitation to participate in OBCS. | 2 months
  Data related to care pathways 2 months after presentation of the DA tool, in both arms: mammograms completed; appointments made to undergo mammography; appointments made to discuss screening; type of professionals contacted by participants (GP, midwife, gynaecologist, other).
Evaluation of the effect of presenting the discutons-mammo.fr DA tool on decisional conflict in subgroups characterized by lower participation in OBCS. | 2 months
  Collection of socio-demographic patient data (home, work, marital status, in receipt of state aid) and health data (long-term illness, history of participation in OBCS, history of participation in colon cancer screening). Data collected 2 months after presentation of the DA tool, in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Rat, M.D. PhD., Study Director — Nantes University Hospital, Faculty of medicine, General Practice Department, Nantes, France; Sandrine Hild, M.D., Principal Investigator — Nantes University Hospital, Faculty of medicine, General Practice Department, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hild S, Teigne D, Ferrat E, Banaszuk AS, Berquet K, Lebon A, Bataille E, Nanin F, Gaultier A, Rat C. Breast cancer: a randomized controlled trial assessing the effect of a decision aid on mammography screening uptake: study protocol. Front Oncol. 2023 Apr 24;13:1128467. doi: 10.3389/fonc.2023.1128467. eCollection 2023. PMID 37168386